CLINICAL TRIAL: NCT06231927
Title: Feasibility and Acceptability of SOLAR Group Program on Decreasing the Distress and Secondary Traumatization of MHPSS Workers After the Earthquake in Türkiye
Brief Title: Feasibility of SOLAR Group Program Among MHPSS Workers After the Earthquake
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ceren Acarturk, Principal Investigator, Koç University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023.371.IRB3.164
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Psychological Distress; Secondary Trauma; Depression; Anxiety
MeSH Terms: conditions — Compassion Fatigue; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): This is an open feasibility trial with single group of individuals receiving the SOLAR intervention program.
  Interventions: Behavioral: The Skills for Life Adjustment and Resilience (SOLAR) program

INTERVENTIONS:
Behavioral: The Skills for Life Adjustment and Resilience (SOLAR) program — The SOLAR program is a 5-session intervention program that aims to introduce participants necessary recovery skills after a traumatic event resulting in a subclinical distress. During the program, participants will be given workbooks including the topics for skill development for recovery and adjustment. At each session, they will discuss these topics with the study coaches.

SUMMARY:
The goal of this intervention program is to provide the feasibility of a culturally adapted version of the SOLAR program among mental health and psychosocial support (MHPSS) workers who provide psychological or psychosocial support to the survivors of the earthquakes on February 6, 2023, in Türkiye. The main questions it aims to answer are:

1. Will the SOLAR Group Program reduce psychological distress at the post-test and follow-up compared to the pre-test?
2. Will the SOLAR Group Program reduce secondary traumatic stress at the post-test and follow-up compared to the pre-test?
3. Will the SOLAR Group Program reduce anxiety and depressive symptoms at the post-test and follow-up compared to pre-test?

Participants will be asked to sign a consent form. Upon accepting it, they will fill out:

* a demographic form,
* the Kessler Psychological Distress Scale (K10),
* Assessment of Suicidal Thoughts for the screening.

Before the SOLAR intervention program, participants will be asked to complete:

* the Secondary Traumatic Stress Scale (STSS),
* Generalized Anxiety Disorder-7 (GAD-7),
* the Patient Health Questionnaire (PHQ-9) if they approve participation in these surveys.

After collecting their pre-test scores, they will receive the SOLAR intervention program. During the program, they will be asked to participate in each session, lasting 5 weeks.

After the program, they will be asked to participate process evaluation interview.

DETAILED DESCRIPTION:
A disaster can be defined as a significant disturbance in the operation and well-being of a community resulting from the convergence of hazardous events with factors such as exposure, and vulnerability. Disasters are grouped into two main categories: natural disasters and technological disasters. Many individuals who survive these disasters face an increased risk of psychological distress and psychopathology, including depressive disorders or Post-Traumatic Stress Disorder (PTSD). PTSD symptoms include intrusion symptoms, avoidance, negative alterations in cognition and mood, arousal and reactivity, or even dissociation. However, as well as being directly exposed to the event, trauma can be indirect by witnessing the event experienced by others and the impact of indirect trauma can be just as significant as that of direct trauma. Family members, friends, neighbours, coworkers, and professionals assisting the primary victims may also undergo similar traumatic symptoms. Many professionals from various fields, such as doctors, nurses, first responders, and mental health workers, are dedicated to helping disaster survivors' short-term and long-term needs. Therefore, they experience similar symptoms of survivors, including re-experiencing the traumatic event, avoidance of reminders of the event, detachment from others, irritability, and persistent arousal like difficulty sleeping. The development of these symptoms due to close contact with the survivor is called secondary traumatic stress (STS). After disasters, it is important to consider the mental health of people who are secondarily exposed to trauma and those who experience the trauma.

Psychological distress refers to an individual's distinct unpleasant emotional state when confronted with a particular stressor, which subsequently damages the person. It is frequently used to describe a wide range of symptoms, including depression and general anxiety symptoms as well as personality traits and behavioral issues. After an exposure to a disaster, many individuals encounter mental health challenges and are more susceptible to developing psychiatric disorders such as anxiety disorders, depressive disorders, and post-traumatic stress disorder (PTSD). These syndromes result in psychological distress and dysfunctionalities in the individual's psychosocial and occupational lives. The symptoms can be seen not only in people who experienced the disaster but also in those who communicated with them. Mental health and psychosocial support (MHPSS) workers face a distinct aspect of their job, which involves being exposed to their clients' experiences of trauma. They introduce interventions in areas such as health, education, abuse and violence, and emergencies to help survivors to deal with the mental health impacts of those experiences. Therefore, MHPSS workers are at risk for developing symptoms of secondary traumatization and psychological distress.

On February 6, 2023, two major earthquakes with magnitudes of 7.7 and 7.6 struck Türkiye and Syria, centered in Kahramanmaraş, Türkiye. Over the course of one month, various numbers of aftershocks continued. This catastrophic event affected approximately 13 million people in 11 Turkish provinces. 50,783 Turkish citizens died and countless individuals lost their loved ones, their homes, and their jobs. This disaster inflicted immense suffering on people in the country, and they had to deal with many major life-changing impacts and issues. The earthquake affected not only the people in the region but also those who went to the region to offer help, and those who observed the unfolding events. Psychosocial support institutions and mental health professionals were some of the ones who went to the region to assist. Interventions should be designed for mental health professionals regarding the secondary traumatization they might encounter in the aftermath of the earthquake.

Skills for Adjustment and Resilience (SOLAR) Program was formed by a team consisting of 21 experts from around the world with expertise in trauma, disaster mental health, and disaster response, representing the USA, UK, Canada, Australia, and Asia. It was designed for the need for practical interventions to address the psychosocial needs of trauma and disaster survivors with subclinical mental health issues. The SOLAR program was intended to be efficient, adaptable in various settings, and easily applicable for trained laypersons and professionals to reach more people with subclinical distress following a traumatic event. It also has a trauma processing unit specifically designed for traumatized individuals. Each session lasts 50 minutes, except for the first session, which is 80 minutes and is delivered face-to-face over five weeks. The SOLAR program was effective in the pilot study with 15 bushfire survivors in Australia (O'Donnell et al., 2020). Furthermore, its effectiveness in reducing depressive and post-traumatic stress symptoms in a group format was also confirmed with 79 people in Tuvalu affected by Tropical Cyclone Pam. Lastly, the program was feasible and useful for improving coping with traumatic events among German trauma survivors with persistent subclinical distress.

This study aims to provide the feasibility of a culturally adapted version of the SOLAR program among MHPSS workers who provide psychological or psychosocial support to the survivors of the earthquakes on February 6, 2023, in Türkiye. As an intervention program, SOLAR aims to examine subclinical distress and adjustment problems following a traumatic experience, in this case, an earthquake. The primary inquiry of this study aimed to assess the feasibility of implementing the SOLAR group program within an open trial among 20 MHPSS workers in the aftermath of a trauma. In addition to the feasibility, the study aims to decrease participants' distress levels as the primary outcome and their secondary traumatization, depression, and anxiety levels as secondary outcomes.

Given the information above, the hypotheses of the current study are as follows:

* The SOLAR Group Program will be feasible and effective among MHPSS workers who have experiences with survivors of the earthquake in Türkiye
* The SOLAR Group Program will reduce psychological distress at the post-test and follow-up compared to the pre-test.
* The SOLAR Group Program will reduce secondary traumatic stress at the post-test and follow-up compared to the pre-test.
* The SOLAR Group Program will reduce anxiety and depressive symptoms at the post-test and follow-up compared to the pre-test.

First, they will receive a consent form for the participation. Upon accepting it, they will fill out a demographic form, the Kessler Psychological Distress Scale (K10) and Assessment of Suicidal Thoughts for the screening. People with scores over 20 on this scale, 18 years of age or above, and MHPSS workers who have no suicidal risk will be included in the study. Before the SOLAR, the intervention program, participants will be asked to complete The Secondary Traumatic Stress Scale (STSS), Generalized Anxiety Disorder-7 (GAD-7), and The Patient Health Questionnaire (PHQ-9) if they approve participation in these surveys. STSS will be used to measure secondary traumatic stress symptoms that they are experiencing. While GAD-7 will be used to measure anxiety, PHQ-9 will be used to measure depression. It will take approximately 20 minutes to attend these surveys. After collecting their pre-test scores, they will receive the SOLAR intervention program.

The SOLAR intervention program was translated and adapted to Turkish by a group of psychologists. Participants will be provided with a workbook that includes topics of the sessions and practice tools of the contents for each session. The content of the workbook includes strategies for maintaining a healthy lifestyle, managing distressing emotions, coming to terms with disaster experiences, getting back to usual activities, and dealing with worry and negative thoughts. The program will be delivered by coaches in weekly sessions for 5 weeks. Each session lasts 50 minutes, except for the first session which is 80 minutes. Coaches will be people who took part in the Turkish adaptation of the program, and they will follow the coach manual. After 5 weeks, post-test scores of the same scales will be assessed. The same scales will be used at the follow-up one month after post-test. There will be no control group in this study.

Since this is a feasibility study, the feasibility outcomes will also be assessed and reported by eligibility rate, recruitment speed, treatment adherence, dropout rate, and process evaluation interview. In this interview, participants will be asked about how they found the intervention in general, how they found the coaches, and their feedback on aspects that could be improved. The informed consent for the process evaluation interview will also be collected from the participants. These interviews will be administered by another researcher other than the coaches conducting the study. The data analysis will be conducted using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* actively working as an MHPSS worker who provides psychosocial support to the survivors of the February 6 earthquake
* having subclinical symptoms of distress (score>20 on The Kessler Psychological Distress Scale (K10)
* no suicidal risk.

Exclusion Criteria:

* not approving the informed consent
* having a suicidal thought.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | 1. approximately a week before intervention for the screening 2. at the end of the intervention 3. one month after the end of the intervention
  The Kessler Psychological Distress Scale (K10)

SECONDARY OUTCOMES:
Secondary traumatic stress | 1. at the beginning of the intervention 2. at the end of the intervention 3. one month after the end of the intervention
  The Secondary Traumatic Stress Scale (STSS)
Depression | 1. at the beginning of the intervention 2. at the end of the intervention 3. one month after the end of the intervention
  The Patient Health Questionnaire (PHQ-9)
Anxiety | 1. at the beginning of the intervention 2. at the end of the intervention 3. one month after the end of the intervention
  Generalized Anxiety Disorder-7 (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Acartürk, Study Director — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Since the data will be collected via Qualtrics, their IP addresses will be available. However, to ensure anonymity in data analysis, participants will be associated with a random identification number or a code to follow data from pre- and post-assessments.
Supporting Information: Study Protocol, ICF
Time Frame: All data will be kept in a locked safe for 10 years. Then, it will be deleted in an untraceable way.
Access Criteria: The researcher and the supervisor of this study will have access to data. As mentioned, participants have different identification numbers or codes.

REFERENCES:
- [Background] O'Donnell ML, Lau W, Fredrickson J, Gibson K, Bryant RA, Bisson J, Burke S, Busuttil W, Coghlan A, Creamer M, Gray D, Greenberg N, McDermott B, McFarlane AC, Monson CM, Phelps A, Ruzek JI, Schnurr PP, Ugsang J, Watson P, Whitton S, Williams R, Cowlishaw S, Forbes D. An Open Label Pilot Study of a Brief Psychosocial Intervention for Disaster and Trauma Survivors. Front Psychiatry. 2020 Jun 26;11:483. doi: 10.3389/fpsyt.2020.00483. eCollection 2020. PMID 32670099